CLINICAL TRIAL: NCT04289883
Title: Nano-particulated and Alginate Whey Protein's Effects on Appetite - Food Structure Approaches Developed Within the StrucSat Project
Brief Title: Food Structure and Satiety
Acronym: StrucSat
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The Covid-19 pandemic that made it impossible to conduct within the timeframe.
Sponsor: Arne Astrup (Other)
Collaborators: University of Copenhagen (Other); Technical University of Denmark (Other); DuPont Nutrition and Health (Industry); Arla Foods (Industry)
Responsible Party: Sponsor-Investigator, Arne Astrup, Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B311
Record Dates: First submitted 2020-02-13; First posted 2020-02-28 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Appetitive Behavior
Keywords: Satiety; Appetite; Food structure
MeSH Terms: conditions — Appetitive Behavior

STUDY DESIGN:
Intervention Model Description: A double-blind, randomised crossover design with four arms divided into two parts.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High molecular weight whey protein-alginate/Calcium alginate (Experimental): Produced from whey protein with different structures (nano-particulated vs. non-particulated whey proteins and high molecular weight whey protein-alginate coacervates vs. calcium alginate) added cream, sucrose and lactose in order for the products to contain all macronutrients and in equal amounts between the intervention and the control products. Additionally, vanilla flavour (Dr. Oetker vanilla extract) is added in order for the test products to taste similar to "koldskål" (a well-known Danish food). All test products will be produced in the dairy pilot plant at Department of Food Science at University of Copenhagen prior to performance of the appetite probe days. All test products will have a pH of 4 and will be manufactured from dry (powdered) ingredients and pasteurized cream. They will be kept refrigerated for a maximum of 3 days prior to use and production will be planned accordingly.
  Interventions: Combination Product: High molecular weight whey protein-alginate coacervates vs calcium alginate (control)
- Nano-particulated whey protein/Non-particulated whey protein (Experimental): Produced from whey protein with different structures (nano-particulated vs. non-particulated whey proteins and high molecular weight whey protein-alginate coacervates vs. calcium alginate) added cream, sucrose and lactose in order for the products to contain all macronutrients and in equal amounts between the intervention and the control products. Additionally, vanilla flavour (Dr. Oetker vanilla extract) is added in order for the test products to taste similar to "koldskål" (a well-known Danish food). All test products will be produced in the dairy pilot plant at Department of Food Science at University of Copenhagen prior to performance of the appetite probe days. All test products will have a pH of 4 and will be manufactured from dry (powdered) ingredients and pasteurized cream. They will be kept refrigerated for a maximum of 3 days prior to use and production will be planned accordingly.
  Interventions: Combination Product: Nano-particulated whey protein vs non-particulated whey protein (control)

INTERVENTIONS:
Combination Product: Nano-particulated whey protein vs non-particulated whey protein (control) — Different particularisations of whey protein were identified to potentially delay digestion based on in vitro studies and to potentially affect appetite and body weight based on animal studies compared to non-particulated whey protein, with nano-particulated whey protein suggested to be more efficient than micro-particulated.
  Arms: Nano-particulated whey protein/Non-particulated whey protein
Combination Product: High molecular weight whey protein-alginate coacervates vs calcium alginate (control) — Different whey protein-alginate coacervates were identified to potentially delay digestion based on in vitro studies and to potentially affect appetite based on animal studies compared to calcium alginate, with high molecular weight alginate suggested to be more efficient than low molecular weight alginate.
  Arms: High molecular weight whey protein-alginate/Calcium alginate

SUMMARY:
Based on in vitro studies identifying changes in food structures potential to delay digestion as well as results from animal studies showing potential of these foods to decrease appetite, nano-particulated whey protein and high molecular weight whey protein-alginate coacervates were chosen to be investigated in humans. Thereby, the aim of this short-term study is to investigate if nano-particulated whey protein has appetite reducing effects in humans compared to non-particulated whey protein (Part 1) as well as if high molecular weight whey protein-alginate coacervates have appetite reducing effects in humans compared to calcium alginate (Part 2).

DETAILED DESCRIPTION:
Based on animal studies in mice, nano-particulated whey protein and high molecular weight whey protein-alginate coacervates are expected to have appetite reducing (and potentially also other) effects, which potentially may be beneficial for body weight management. In order to investigate these effects in humans, this study is divided into two parts (Part 1 and Part 2), of which the specific objectives are specified below:

Part 1: The objective of this part of the study is to examine if nano-particulated whey protein can reduce appetite compared with non-particulated whey protein.

Part 2: The objective of this part of the study is to examine if high molecular weight whey protein-alginate coacervates can reduce appetite compared to calcium alginate.

A double-blind, randomised crossover design with four arms divided into the two parts will be applied. After having successfully completed screening procedures, eligible participants will be invited to two separate appetite probe days with particulated whey protein followed by at least 14 days break followed by another two separate appetite probe days with the whey protein-alginate coacervates. The appetite probe days must be separated by at least 7 days, but there is no upper limit for days in between, as long as the participants remain weight stable and do not change diet or physical activity level significantly. The study includes a total of five visits to the study site.

For standardisation, 48 hours before the appetite probe days, the participants will be asked to consume a regular diet compliant to what they usually eat and no excessive alcohol consumption (not above 5 units and no alcohol at all from 8 pm the night before the appetite probe days) or intense physical activity is allowed. Within each part of the study, the participants will be instructed to consume similar meals the evening before the appetite probe days and the meal must be consumed at approximately the same time. The participants will also be instructed to go to bed at the same time in the evening prior to the appetite probe days. Additionally, the participants must arrive at the study facilities in the morning after an overnight fast (from 10 pm) using non strenuous means of transportation. Furthermore, over the course of the study (from screening (visit 1) to completion of the last appetite probe day (visit 5)), the participants are not allowed to change body weight (±3 kg), diet or physical activity level (as judged by the sub-investigator). The participants will be weighed and asked about compliance with additional standardisation criteria in a room away from the other participants before initiating each appetite probe day. Possible non-compliance with the standardisation will be judged whether to result in re-scheduling of the visit or to be recorded as a protocol deviation.

Participants arrive at the study facility in the morning. Compliance with standardisation is controlled along with registration of possible adverse events and use of concomitant medications. During the appetite probe days, participants are settled together in an open office, where they are separated at individual tables. During the ad libitum lunch, participants are settled into individual feeding cubicles, where they cannot see each other and are instructed not to talk to each other.

VAS' will be completed for measurement of fasting levels of self-reported appetite.

The test products will be provided as a standardised fixed breakfast and as a standardised fixed mid-morning meal provided 3 hour and 1 hour prior to the ad libitum lunch, respectively.

Immediately before and after the test products and the ad libitum lunch and at 30 minutes intervals, VAS' will be completed assessing self-reported appetite.

After the ad libitum lunch, the participants will be free to leave the laboratory. They will be provided with a snack box including a variety of foods to including a ready-to-heat dish for dinner etc. providing approximately 10000 kJ. The participants will be instructed only to consume foods and drinks (water excepted) from the snack box for the remaining of the days, and to be focussed while eating and only eat until feeling comfortably full. The participants will be instructed to complete a diary registering the time point of consumption of which items from the snack box (and potential additional items). If consuming any foods or energy containing drinks besides those provided in the snack box, the participants will be instructed to register the type and amount consumed. Within the diary, the participants will also be instructed to register the time of going to bed on the day of the appetite probe day. At the second appetite probe day within each part of the study, the participants will be instructed to go to bed at approximately the same time as registered at the first appetite probe day within each part of the study. On the following day after each appetite probe day, the participants will be instructed to hand in the leftovers from the snack box and the diary at the research facility.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have provided written informed consent
* Healthy men and women (at least 40% of each gender)
* Age between 18 and 45 years
* BMI between 22.0-30.0 kg/m2
* Regular breakfast eaters (eating breakfast ≥ 4 times a week)

Exclusion Criteria:

* Participants unable to consume the test products (the test product will be presented at screening)
* Participants not able to comply with the study protocol, including consumption of the specific study foods served during lunch and in the snack box (the study foods will be presented at screening)
* Any known food allergies or food intolerance likely to affect the present study
* Significant health problems as judged by the principal investigator
* Taking any medication or supplements known to affect appetite or body weight within the past month and/or during the study, as judged by the principal investigator
* Smoking, smoking cessation within the past 3 months or nicotine use (electronic cigarettes, gum etc.). Irregular smokers accepted
* Self-reporting currently dieting or having lost/gained significant amount of weight (±3 kg) in the previous 3 months
* Significant weight changes (±3 kg) over the course of the study (from screening to completion of last appetite probe day)
* Significant changes in physical activity patterns in the past 4 weeks or significant changes over the course of the study (from screening to completion of last appetite probe day), as judged by the sub-investigator
* Significant changes in diet in the past 4 weeks or significant changes over the course of the study (from screening to completion of last appetite probe day) as judged by the sub-investigator
* Participants who work in appetite related areas
* Simultaneous or within the past month participating in other clinical trials that can interfere with the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-reporting
Enrollment: 0 (Actual)
Dates: Start 2020-04-25 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
24-hour energy intake (kJ) | 24 hour
  Difference in 24-hour energy intake (the total energy intake from the test products, the ad libitum lunch and the ad libitum snack box) between exposure to the experimental conditions compared to the matching control conditions.

SECONDARY OUTCOMES:
Energy intake (kJ) at each of the ad libitum meals | Lunch: 30 minutes; Snack box: from 12.00 pm until going to bed (app. 11 hour)
  Difference in energy intake at each of the ad libitum meals (lunch and snack box) between exposure to the experimental conditions compared to the matching control conditions.
Visual analogue scales (VAS) of self-reported appetite assessed throughout the appetite probe days while being in the laboratory | 3 hour
  Difference in perceptions of satiety, fullness, hunger and predicted prospective food consumption between exposure to the experimental conditions compared to the matching control conditions using VAS (0-100 mm with 0 indicating no hunger or perccieved ability to consume food / no satiety or no fullness).
Satiety quotient (SQ) | 30 minutes
  Difference in SQ between exposure to the experimental conditions compared to the matching control conditions is assessed by analysing the VAS assessments before and after the ad libitum lunch in relation to the energy consumed at the test meal will be assessed.
Visual analogue scales of self-reported nausea and well-being assessed throughout the appetite probe days while being in the laboratory | 3 hour
  Difference in perceptions of nausea and well-being between exposure to the experimental conditions compared to the matching control conditions using VAS (0-100 mm with 0 indicating no nausea).
Visual analogue scales of self-reported product palatability | 5 minutes (assessed after both exposures at each appetite probe day)
  Difference in perceptions of palatability of the test products between exposure to the experimental conditions compared to the matching control conditions using VAS (0-100 mm with 0 indicating low palatability of the product).

CONTACTS AND LOCATIONS:
Overall Officials: Anders Sjödin, PhD, Principal Investigator — University of Copenhagen, Department of Nutrition, Exercise and Sports
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen, Copenhagen, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared